CLINICAL TRIAL: NCT01796587
Title: Non-Interventional Study Among Users Of LoFric Origo
Status: Completed | Type: Observational
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: LOF-0017
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Intermittent Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LoFric Origo
  Interventions: Device: LoFric Origo

INTERVENTIONS:
Device: LoFric Origo

SUMMARY:
Primary objective: To evaluate compliance of LoFric Origo in a general intermittent catheterization (IC) population with the use of LoFric Origo, by means of a subjective assessment scale

Secondary objectives:

* To evaluate the subject's perception associated with the use of the LoFric Origo, by means of a subjective assessment scale
* To evaluate the subject's discomfort associated with the use of the LoFric Origo, by means of a subjective assessment scale
* To observe and collect data on bladder regimen/IC frequency by assessments of descriptive data of demography, catheter therapy, history and other patient reported outcomes.

Study Design: Non-interventional study, multicentre, prospective study. Target Subject Population: General intermittent catheterization, LoFric Origo male users.

Medical Device: LoFric Origo

Study Variable(s):

* Primary variable: Use or No use of LoFric Origo after 8 weeks.
* Secondary variable(s): patient reported questionnaire with regards to perception, discomfort, diagnose, health status, catheter history and other patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Males, aged 18 years and over
3. Practice intermittent self-catheterization, at least one time daily
4. Subjects using LoFric Origo
5. Able to read and fill out a patient reported questionnaire as judge by the investigator
6. The prescription of/decision to use the medical device is separated from the decision to include the subject in the study.

Exclusion Criteria

1. Simultaneous participation in any interfering clinical study
2. On-going, symptomatic urinary tract infection (UTI) at enrolment as judged by the investigator
3. Involvement in the planning and/or conduct of the study (applies to both Wellspect HealthCare staff and staff at the study site)
4. Previous enrolment in the present study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed LoFric Origo for intermittent catheterization, attending any of the involved clinics.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects still using LoFric Origo | 8 weeks
  Outcome variable is to measure the proportion of subjects still using LoFric Origo after 8 weeks through subjective assessment scales.

SECONDARY OUTCOMES:
Perception of LoFric Origo | 8 weeks
  Perception is a subjective sensation/impression which may be expressed in different ways. The concept of Perception, in this observational study, reflects each subject's own experience when using LoFric Origo and the subjects will evaluate the catheters with respect to a number of predetermined variables.
Discomfort | 8 weeks
  Evaluate subject's perceived discomfort associated with the use of the LoFric Origo, in terms of pain, burning sensation, bleeding and other discomfort.

CONTACTS AND LOCATIONS:
Locations (19):
- Belgium (3):
  - Centre de Traumatologie et de Readaptation, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Domaine Universitaire du Sart Tilman, Liége
- France (4):
  - Groupe Urologique de la Clinique Saint Augustin, Cabinet de Neuro-Urologie, Bordeaux
  - Hôpital Raymond Poincaré, Service de Neuro-Urologie, Urologie et Sexologie, Garche
  - Hôpital Tenon, Service de Neuro-Urologie et Explorations Périnéales, Paris
  - Hôpital Henry Gabrielle, Unité A1 - Service de Rééducation Périnéale et Sexologique, Saint-Genis-Laval
- Netherlands (2):
  - Rivas Zorggroep, Gorinchem, South Holland
  - U.M.C. St. Radboud, Nijmegen
- Norway (4):
  - Akershus Universitetssykehus HF Urologisk poliklinikk, Lørenskog
  - Sunnaas Sykehus HF Urodynamisk laboratorium, Nesoddtangen
  - Oslo Universitetssykehus HF - Rikshospitalet Urologisk poliklinikk, Oslo
  - Stavanger Universitetssjukehus, Urologisk poliklinikk, Stavanger
- Switzerland (2):
  - Schweizer Paraplegiker-Zentrum, Neuro-Urologie, Nottwil
  - Clinique romande de réadaptation, Sion
- United Kingdom (4):
  - University Hospitals Coventry and Warwickshire NHS Trust Walsgrave Hospital, Coventry, Coventry
  - Musgrove Park Hospital, Taunton, Somerset
  - Exeter RD&E Hospital, Exeter
  - National Hospital for Neurology and Neurosurgery Queens Square, London